CLINICAL TRIAL: NCT00748189
Title: A Phase III, Open Label, Randomized, Multicenter Trial of Ofatumumab Added to Chlorambucil Versus Chlorambucil Monotherapy in Previously Untreated Patients With Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab + Chlorambucil vs Chlorambucil Monotherapy in Previously Untreated Patients With Chronic Lymphocytic Leukemia
Acronym: COMPLEMENT 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Majority of patients (62%) had been treated with next line therapies, including new highly effective therapies confounding the interpretation of the OS results.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: OMB110911; OMB110911 (Other: Novartis)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: Safety; Untreated; Efficacy; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia (CLL), untreated; Ofatumumab; Oncology
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — Chlorambucil; Tablets; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ofatumumab + chlorambucil (Experimental): ofatumumab dose: cycle 1 300mg day 1 and 1000mg day 8, subsequent cycles: 1000mg at day 1 every 28 days; chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 treatment cycles
  Interventions: Drug: chlorambucil, tablets; Drug: ofatumumab (GSK1841157) infusion
- chlorambucil (Active Comparator): chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 cycles
  Interventions: Drug: chlorambucil, tablets

INTERVENTIONS:
Drug: chlorambucil, tablets — 2mg tablets, chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 cycles
Drug: ofatumumab (GSK1841157) infusion — iv infusion; dose: cycle 1 300mg day 1 and 1000mg day 8, subsequent cycles: 1000mg at day 1 every 28 days;
  Other Names: chlorambucil; tablets
  Arms: ofatumumab + chlorambucil

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ofatumumab added to chlorambucil in patients with untreated Chronic Lymphocytic Leukemia.

DETAILED DESCRIPTION:
Chlorambucil, is currently approved for treatment of frontline chronic lymphocytic leukemia, especially, but not limited to the ailing and elderly patient population. Several other more aggressive treatment options are available (e.g. fludarabine), however they are not suitable for all CLL patients, especially the ailing and elderly, due to greater toxicity. Ofatumumab is effective with low toxicity. The addition of ofatumumab to chlorambucil offers potentially a more effective therapy, with limited toxicity. The objective of this study was to evaluate progression-free survival (PFS), overall response and overall survival in subjects with previously untreated CLL with ofatumumab added to chlorambucil versus chlorambucil.

ELIGIBILITY:
Inclusion Criteria:

* confirmed CLL diagnosis and active CLL requiring treatment
* considered inappropriate for fludarabine-based therapy
* not been treated for CLL before
* fully active at a minimum or fully capable of selfcare and up and about more than 50% of waking hours
* age 18yrs or older
* signed written informed consent

Exclusion Criteria:

* prior CLL therapy
* abnormal/inadequate blood values, liver, and kidney function
* certain heart problems, active or chronic infections, serious significant diseases, active autoimmune hemolytic anemia (AIHA) requiring treatment, other current cancer or within last 5 years
* CLL transformation
* CLL central nervous system involvement
* current participation in other clinical study
* inability to comply with the protocol activities
* lactating or pregnant women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2008-12-22 (Actual); Primary Completion 2013-03-20 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (140):
- United States (28):
  - Novartis Investigative Site, Sedona, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Murrieta, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, New Port Richey, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Ocoee, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Lee's Summit, Missouri
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Midland, Texas
  - Novartis Investigative Site, Odessa, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Vancouver, Washington
  - Novartis Investigative Site, Yakima, Washington
- Belgium (5):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Pierre-Bénite
- Germany (17):
  - Novartis Investigative Site, Karlsruhe, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Lehrte, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Moenchengladbach-Rheydt, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Saarbrücken, Saarland
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- India (5):
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Pune
- Ireland (7):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, James Street
  - Novartis Investigative Site, Limerick
  - Novartis Investigative Site, Tullamore
  - Novartis Investigative Site, Waterford
- Italy (13):
  - Novartis Investigative Site, Bari, Apulia
  - Novartis Investigative Site, Potenza, Basilicate
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Albano Laziale (Roma), Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Brescia, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Palermo, Sicily
  - Novartis Investigative Site, Ascoli Piceno, The Marches
  - Novartis Investigative Site, Venezia - Mestre, Veneto
  - Novartis Investigative Site, Vicenza, Veneto
  - Novartis Investigative Site, Udine
- Netherlands (6):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, The Hague
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- Spain (5):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Hospitalet de Llobregat (Barcelona)
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Sweden (3):
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (29):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Sunderland, Tyne
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, Carshalton
  - Novartis Investigative Site, Cornwall
  - Novartis Investigative Site, Dudley
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Milton Keynes
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Peterborough
  - Novartis Investigative Site, Rhyl, Denbighshire
  - Novartis Investigative Site, Salford
  - Novartis Investigative Site, Stoke-on-Trent
  - Novartis Investigative Site, Swindon
  - Novartis Investigative Site, Uxbridge

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tausch E, Beck P, Schlenk RF, Jebaraj BJ, Dolnik A, Yosifov DY, Hillmen P, Offner F, Janssens A, Babu GK, Grosicki S, Mayer J, Panagiotidis P, McKeown A, Gupta IV, Skorupa A, Pallaud C, Bullinger L, Mertens D, Dohner H, Stilgenbauer S. Prognostic and predictive role of gene mutations in chronic lymphocytic leukemia: results from the pivotal phase III study COMPLEMENT1. Haematologica. 2020 Oct 1;105(10):2440-2447. doi: 10.3324/haematol.2019.229161. PMID 33054084
- [Derived] Hillmen P, Robak T, Janssens A, Babu KG, Kloczko J, Grosicki S, Doubek M, Panagiotidis P, Kimby E, Schuh A, Pettitt AR, Boyd T, Montillo M, Gupta IV, Wright O, Dixon I, Carey JL, Chang CN, Lisby S, McKeown A, Offner F; COMPLEMENT 1 Study Investigators. Chlorambucil plus ofatumumab versus chlorambucil alone in previously untreated patients with chronic lymphocytic leukaemia (COMPLEMENT 1): a randomised, multicentre, open-label phase 3 trial. Lancet. 2015 May 9;385(9980):1873-83. doi: 10.1016/S0140-6736(15)60027-7. Epub 2015 Apr 14. PMID 25882396
- [Derived] Jewell RC, Laubscher K, Lewis E, Fang L, Gafoor Z, Carey J, McKeown A, West S, Wright O, Sedoti D, Dixon I, Hottenstein CS, Chan G. Assessment of the effect of ofatumumab on cardiac repolarization. J Clin Pharmacol. 2015 Jan;55(1):114-21. doi: 10.1002/jcph.376. Epub 2014 Aug 21. PMID 25103870

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) were stratified by age (<65 years vs. >=65years), stage (Binet A vs. B vs. C) and Eastern Cooperative Oncology Group (ECOG) performance status (0-1 vs. 2). Participants in each stratum were then centrally randomized in a 1:1 ratio to receive ofatumumab plus chlorambucil (O+CHL) or chlorambucil alone (CHL).
Groups:
- Chlorambucil: Participants with previously untreated chronic lymphocytic leukemia (CLL) received chlorambucil monotherapy 10 milligram (mg)/meter squared (m^2) orally on Days 1-7 of every 28-day cycle for a minimum of 3 cycles until best response or a maximum of 12 cycles.
- Ofatumumab + Chlorambucil: Participants with CLL received intravenous (IV) infusions of ofatumumab on Day 1 (300 mg) and Day 8 (1000 mg) in the first cycle, followed by IV infusions of 1000 mg on the first day of each subsequent 28-day cycle in combination with chlorambucil 10 mg/m^2 orally on Days 1-7 of every 28-day cycle for a minimum of 3 cycles until best response or a maximum of 12 cycles.
Period: Overall Study
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Started | 226 | 221
Completed | 10 | 9
Not Completed | 216 | 212
Not completed — Death | 99 | 84
Not completed — Withdrawal by Subject | 23 | 29
Not completed — Physician Decision | 16 | 5
Not completed — Lost to Follow-up | 8 | 15
Not completed — Study terminated by Sponsor | 70 | 79

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomized subjects regardless of whether or not they received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil | Total
Number analyzed (Participants) | 226 | 221 | 447
Age, Customized [Median (Full Range); unit: Years]
  Years | 70 [36 to 91] | 69 [35 to 92] | 69 [35 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 79 | 165
  Male | 140 | 142 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 2 | 4 | 6
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 22 | 19 | 41
  Asian - Mixed Race | 0 | 2 | 2
  White | 201 | 196 | 397

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), as Assessed by the Independent Review Committee (IRC)
Description: PFS is defined as the interval of time between the date of randomization and the earlier of the date of disease progression (PD) and the date of death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlarged lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Par. who were alive and had not progressed at the time of analysis or if a progression event or death occurred after extensive lost-to-follow-up time or if new anti-cancer therapy was started were censored at the date of the last visit with adequate assessment.
Time Frame: From randomization to the date of first documented disease progression or death due to any cause, whichever occured first, reported between day of first patient randomized up to about 49 months
Population: Intent-to-Treat (ITT) Population: all par. randomized to study treatment regardless of whether or not they received treatment. PFS was assessed by a blinded independent review committee according to the International Workshop for Chronic Lymphocytic Leukemia (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Months | 13.1 [10.6 to 13.8] | 22.4 [19.0 to 25.2]
Statistical Analysis 1: Comparison: Chlorambucil vs Ofatumumab + Chlorambucil; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.45 to 0.72] — Hazard ratios are obtained using the Pike estimator

2. Secondary Outcome: Number of Participants With the Best Overall Response (OR), as Assessed by the IRC
Description: OR is defined as the number of participants achieving an objective response (complete response [CR], CR with incomplete bone marrow recovery [CRi], partial response [PR], and nodular PR [nPR]). CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
Time Frame: From randomization until the 259th PFS event occurred, up to about 49 months
Population: ITT population. Only those participants with data available at the indicated time points were analyzed. OR was according to the International Workshop for Chronic Lymphocytic Leukemia (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines. The 95% exact binomial confidence interval is for CR+CRi+nPR+PR.
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Participants
  CR | 3 | 27
  CRi | 0 | 5
  nPR | 0 | 1
  PR | 152 | 149

3. Secondary Outcome: Number of Participants Who Were Negative for Minimal Residual Disease (MRD)
Description: MRD was performed by flow cytometry on a bone marrow or peripheral blood sample taken at least 2 months after final treatment. MRD negative was defined as less than one CLL cell per 10000 leukocytes.
Time Frame: From randomization until the 259th PFS event occurred (Median follow-up approximately 28.9 months)
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Participants
  MRD negative, irrespective of response | 8 | 26
  MRD negative, with an IRC-assessed CR | 0 | 10

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death due to any cause. Each participant was followed at the time when the total IRC-assessed PFS events occurred. Participants who had not died were censored at the date of last contact.
Time Frame: From randomization up to about 111 months
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Months | 84.67 [74.25 to NA] — the upper limit of the confidence interval was not estimable due to insufficient number of patients with events. | NA [84.50 to NA] — the median/upper limit of the confidence interval was not estimable due to insufficient number of patients with events.
Statistical Analysis 1: Comparison: Chlorambucil vs Ofatumumab + Chlorambucil; Test type: Other; p = 0.363, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.65 to 1.17] — hazard ratios are obtained using the Pike estimator. A hazard ratio <1 indicates a lower risk with O+CHL treatment compared with chlorambucil

5. Secondary Outcome: Time to Response, as Assessed by the IRC
Description: Time to response is defined as the time from randomization to the first response (CR, CRi, nPR, or PR). CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM. Participants with unknown or missing responses were considered as non-responders. Only responders (CR, CRi, PR, nPR) were included in the analysis.
Time Frame: From randomization uo to about 27 months
Population: ITT population. Time to response was measured using the International Workshop for CLL (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines 2008.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 154 | 182
Months | 1.9 [1.2 to 1.9] | 1.2 [1.0 to 1.9]

6. Secondary Outcome: Duration of Response (DOR), as Assessed by the IRC
Description: DOR is defined as the time from the initial response (CR, CRi, nPR, or PR) to the first documented sign of PD or death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlarged lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Par. who were alive and had not progressed at the time of analysis or if a progression event occurred after extensive lost-to-follow-up time (>= 12 weeks) were censored at the date of the last visit with adequate assessment. Par. with unknown or missing responses were considered as non-responders.
Time Frame: From randomization up to about 43 months
Population: ITT population. Only those participants with data available at the indicated time points were analyzed. Only responders (CR, CRi, PR, nPR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 154 | 182
Months | 13.2 [10.8 to 16.4] | 22.1 [19.1 to 24.6]

7. Secondary Outcome: Time to Progression, as Assessed by the IRC
Description: Time to progression is defined as the time from the date of randomization to disease progression (PD). PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlarged lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Participants who were alive and had not progressed at the time of analysis or if a progression event occurred after extensive lost-to-follow-up time were censored at the date of the last visit with adequate assessment.
Time Frame: From randomization up to about 49 months
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Months | 13.6 [11.2 to 14.6] | 23.1 [21.2 to 25.8]

8. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy is defined as the time from randomization until the start of the next-line of treatment.
Time Frame: From randomization up to about 49 months
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 99 | 64
Months | 24.67 [22.57 to 29.08] | 39.82 [34.69 to 48.79]

9. Secondary Outcome: Number of Participants With Improvement in ECOG Performance Status of 0 or 1
Description: The ECOG performance status scales and criteria are used by doctors and researchers to assess how a participant's disease is progressing, how the disease affects the daily living, and determines appropriate treatment and prognosis. Grade 0, fully active, able to carry on all pre-disease performance without restriction. Grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about more than 50% of waking hours. Grade 3, capable of only limited selfcare; confined to bed or chair more than 50% of waking hours. Grade 4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. Grade 5, dead. Participants with an ECOG performance status of 0 or 1 are shown..
Time Frame: Baseline, Cycle 3 Day 1, 1 month Follow-up
Population: ITT population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants
  ECOG (0, 1) at Baseline: number analyzed (Participants) | 226 | 217
  ECOG (0, 1) at Baseline | 209 | 200
  ECOG (0, 1) at Cycle 3 Day 1: number analyzed (Participants) | 199 | 196
  ECOG (0, 1) at Cycle 3 Day 1 | 184 | 189
  ECOG (0, 1) 1 Month Follow-up: number analyzed (Participants) | 196 | 199
  ECOG (0, 1) 1 Month Follow-up | 183 | 191

10. Secondary Outcome: Number of Participants With Improvement in Constitutional Symptoms (CS)
Description: Assessment for the presence of the following symptoms were performed at Screening, Day 1 of each treatment cycle and at every Follow-up visit: night sweats (without signs of infection); unexplained, unintentional weight loss >= 10% within the previous 6 months; recurrent, unexplained fever of greater than 38 degrees celsius or 100.5 degrees fahrenheit for 2 weeks; and extreme fatigue. The best response refers to overall best response in terms of CR, CRi, PR or nPR. Data are presented for constitutional response= yes and no.
Time Frame: Baseline, Cycle 3 Day 1, and 1 month Follow-up
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Participants
  CS present, Baseline, n=226, 221 | 120 | 118
  CS present, Cycle 3 Day 1, n=198, 199: number analyzed (Participants) | 198 | 199
  CS present, Cycle 3 Day 1, n=198, 199 | 44 | 33
  CS present, 1 Month Follow-up, n=198, 200: number analyzed (Participants) | 198 | 200
  CS present, 1 Month Follow-up, n=198, 200 | 23 | 22

11. Secondary Outcome: Number of Participants With a Human Anti-human Antibody (HAHA) Positive Result
Description: Serum samples for analysis of HAHA were collected at Baseline (Screening), Cycle 4 Day 1 (after 3 months of treatment), and at 1 month and 6 months post last dose of ofatumumab. All samples were first tested in a screening step; positive samples from the screening were further evaluated in a confirmation test. The confirmed positive samples were reported as HAHA-positive and further evaluated in the titration test to obtain a titer of HAHA.
Time Frame: Baseline, Cycle 4 Day 1, 1 Month Follow-up, and 6 Month Follow-up
Population: Safety population: all participants who received at least 1 dose of a study drug. Only participants with post-ofatumumab HAHA Results are included.
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 217
Participants |  | 0

12. Secondary Outcome: Cmax and Ctrough of Ofatumumab
Description: Blood samples were collected to assess the plasma concentration of ofatumumab. Maximum concentration (Cmax) and observed drug concentration prior to the next dose (Ctrough) were determined. Blood samples were collected from participants who received ofatumumab plus chlorambucil at pre-dose and 0.5 hours after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, pre-dose samples were collected prior to ofatumumab administration at Cycles 2, 3, 5, 6, 9 and 12 (Days 29, 57, 113, 141, 225 and 309), depending on the duration of treatment.
Time Frame: Cycle 1 Day 1,Cycle 1 Day 8, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, and Cycle 9 Day 1
Population: Pharmacokinetic (PK) Population: all participants for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms/Milliliter (µg/mL)
Groups:
- Chlorambucil: Participants with previously untreated chronic lymphocytic leukemia (CLL) received chlorambucil monotherapy 10 milligram (mg)/meter squared (m^2) orally on Days 1-7 of every 28-day cycle for up to 12 cycles.
- Ofatumumab + Chlorambucil: Participants with CLL received intravenous (IV) infusions of ofatumumab on Day 1 (300 mg) and Day 8 (1000 mg) in the first cycle, followed by IV infusions of 1000 mg on the first day of each subsequent 28-day cycle up to 12 cycles in combination with chlorambucil 10 mg/m^2 orally on Days 1-7 of every 28-day cycle for up to 12 cycles.
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 193
Micrograms/Milliliter (µg/mL)
  Cmax, Cycle 1 Day 1, n=0, 176: number analyzed (Participants) | 0 | 176
  Cmax, Cycle 1 Day 1, n=0, 176 |  | 51.8 (1.03)
  Cmax, Cycle 1 Day 8, n=0, 193 |  | 241 (0.46)
  Cmax, Cycle 4 Day 1, n=0, 169: number analyzed (Participants) | 0 | 169
  Cmax, Cycle 4 Day 1, n=0, 169 |  | 285 (0.44)
  Ctrough, Cycle 1 Day 8, n=0, 99: number analyzed (Participants) | 0 | 99
  Ctrough, Cycle 1 Day 8, n=0, 99 |  | 2.5 (5.85)
  Ctrough, Cycle 2 Day 1, n=0, 138: number analyzed (Participants) | 0 | 138
  Ctrough, Cycle 2 Day 1, n=0, 138 |  | 5.2 (15.37)
  Ctrough, Cycle 3 Day 1, n=0, 142: number analyzed (Participants) | 0 | 142
  Ctrough, Cycle 3 Day 1, n=0, 142 |  | 6.2 (17.06)
  Ctrough, Cycle 4 Day 1, n=0, 147: number analyzed (Participants) | 0 | 147
  Ctrough, Cycle 4 Day 1, n=0, 147 |  | 15.5 (7.99)
  Ctrough, Cycle 5 Day 1, n=0, 149: number analyzed (Participants) | 0 | 149
  Ctrough, Cycle 5 Day 1, n=0, 149 |  | 33.5 (3.61)
  Ctrough, Cycle 6 Day 1, n=0, 155: number analyzed (Participants) | 0 | 155
  Ctrough, Cycle 6 Day 1, n=0, 155 |  | 45.9 (2.77)
  Ctrough, Cycle 9 Day 1, n=0, 56: number analyzed (Participants) | 0 | 56
  Ctrough, Cycle 9 Day 1, n=0, 56 |  | 55.6 (3.50)

13. Secondary Outcome: Total Plasma Clearance (CL) of Ofatumumab
Description: Plasma clearance is defined as the plasma volume which is totally cleared of drug per unit of time. Blood samples were collected from participants who received ofatumumab plus chlorambucil at pre-dose and 0.5 hours after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, pre-dose samples were collected prior to the ofatumumab administration at Cycles 2, 3, 5, 6, 9 and 12 (Days 29, 57, 113, 141, 225 and 309), depending on duration of treatment. Samples were also collected during clinic visits on Day 15 (during Cycle 1) and Day 43 (during Cycle 2) and at 1, 3, and 6 months post-treatment.
Time Frame: Cycle 4 Day 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter/hour (mL/h)
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 183
Milliliter/hour (mL/h) |  | 15.4 (0.73)

14. Secondary Outcome: AUC(0-tau) of Ofatumumab
Description: Area under the concentration time curve over the dosing interval [AUC(0-tau)] is a measure of drug exposure over time. AUC(0-tau) is defined as the area under the ofatumumab plasma concentration-time curve from dosing to time tau, where tau is the length of the dosing interval of ofatumumab. For estimation of AUC(0-tau), blood samples were collected from participants who received ofatumumab plus chlorambucil at pre-dose and 0.5 hous after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, pre-dose samples were collected prior to the ofatumumab administration at Cycles 2, 3, 5, 6, 9 and 12 (Days 29, 57, 113, 141, 225 and 309), depending on duration of treatment. Samples were also collected during clinic visits on Day 15 (during Cycle 1) and Day 43 (during Cycle 2) and at 1, 3, and 6 months post-treatment.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 4 Day 1
Population: PK Population. Only those participants available at the indicated time points were assessed. The number of participants assessed at each time point is indicated by "n=X,X.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg x hours/mL
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 208
µg x hours/mL
  Cycle 1 Day 1, n=0, 193: number analyzed (Participants) | 0 | 193
  Cycle 1 Day 1, n=0, 193 |  | 2621 (0.76)
  Cycle 1 Day 8, n=0, 208 |  | 25369 (0.87)
  Cycle 4 Day 1, n=0, 183: number analyzed (Participants) | 0 | 183
  Cycle 4 Day 1, n=0, 183 |  | 65100 (0.73)

15. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ofatumumab
Description: Volume of distribution at steady state (Vss) is defined as the distribution of a drug between plasma and the rest of the body at steady state. Blood samples were collected from participants who received ofatumumab plus chlorambucil at predose and 0.5 hour after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, pre-dose samples were collected prior to ofatumumab administration at Cycles 2, 3, 5, 6, 9 and 12 (Days 29, 57, 113, 141, 225 and 309), depending on the duration of the treatment. Samples were also collected during clinic visits on Day 15 (during Cycle 1) and Day 43 (during Cycle 2) and at 1, 3, and 6 months post-treatment.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 4 Day 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 208
Liters
  Vss, Cycle 1 Day 1, n=0, 193: number analyzed (Participants) | 0 | 193
  Vss, Cycle 1 Day 1, n=0, 193 |  | 7.78 (0.55)
  Vss, Cycle 1 Day 8, n=0, 208 |  | 7.77 (0.54)
  Vss, Cycle 4 Day 1, n=0, 183: number analyzed (Participants) | 0 | 183
  Vss, Cycle 4 Day 1, n=0, 183 |  | 8.06 (0.53)

16. Secondary Outcome: Plasma Half Life (t1/2) of Ofatumumab
Description: The terminal half-life (t1/2) of ofatumumab is defined as the time required for the plasma concentration of ofatumumab to reach half of its original concentration. Blood samples were collected to assess the plasma half-life of ofatumumab. Blood samples were collected from participants who received ofatumumab plus chlorambucil pre-dose and 0.5 hours after the end of the ofatumumab infusion at treatment Cycle 1 and Cycle 4 (Days 1, 8, and 85). In addition, pre-dose samples were collected prior to ofatumumab administration at Cycles 2, 3, 5, 6, 9 and 12 (Days 29, 57, 113, 141, 225 and 309), depending on the duration of the treatment. Samples were also collected during clinic visits on Day 15 (during Cycle 1) and Day 43 (during Cycle 2) and at 1, 3, and 6 months post-treatment.
Time Frame: Cycle 4 Day 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 0 | 183
hours |  | 445 (1.05)

17. Secondary Outcome: Dose-normalized Cmax of Chlorambucil and Phenylacetic Acid Mustard (PAAM)
Description: Blood samples for the determination of serum concentrations of chlorambucil and its metabolite PAAM were collected from participants in a substudy on Cycle 3 Day 1. The maximum observed concentration (Cmax) of chlorambucil and PAAM normalized to the administered dose was determined as a measure of exposure and compared to reference data from a prior study (LEUA1001) [No NCT number available for this study; GlaxoSmithKline Document Number RM1998/00449/00].
Time Frame: Cycle 3 Day 1
Population: Chlorambucil/PAAM pharmacokinetic (PK) Population (substudy): all participants for whom a chlorambucil/PAAM sample is obtained and analyzed.
Measure: Geometric Mean (Standard Deviation); unit: nanograms per milliliter per milligram
Groups:
- Study OMB110911: Ofatumumab + Chlorambucil: Participants with CLL received intravenous (IV) infusions of ofatumumab on Day 1 (300 mg) and Day 8 (1000 mg) in the first cycle, followed by IV infusions of 1000 mg on the first day of each subsequent 28-day cycle in combination with chlorambucil 10 mg/m^2 orally on Days 1-7 of every 28-day cycle for a minimum of 3 cycles until best response or a maximum of 12 cycles.
- Study LEUA1001: Chlorambucil: Participants with CLL, Non-Hodgkin's lymphoma or other refractory malignancies received three different formulations of a 0.2 mg/kilogram(kg) chlorambucil tablet orally with a two-day interval between drug administration.
Arm/Group | Study OMB110911: Ofatumumab + Chlorambucil | Study LEUA1001: Chlorambucil
Number analyzed (Participants) | 7 | 12
nanograms per milliliter per milligram
  Chlorambucil Cmax/Dose | 27.1 (0.32) | 38.4 (0.36)
  PAAM Cmax/Dose | 19.3 (0.23) | 24.3 (0.30)
Statistical Analysis 1: Comparison: Study OMB110911: Ofatumumab + Chlorambucil vs Study LEUA1001: Chlorambucil; Test type: Non-Inferiority or Equivalence — Comparability of dose-normalized chlorambucil Cmax values with ofatumumab in current study and without ofatumumab in prior study; Ratio of Cmax/Dose = 0.71, 90% CI 2-sided [0.53 to 0.94] — Ratio of Cmax/Dose is the ratio of dose-normalized chlorambucil Cmax values when given with ofatumumab in the current study and without ofatumumab in the prior study (LEUA1001)
Statistical Analysis 2: Comparison: Study OMB110911: Ofatumumab + Chlorambucil vs Study LEUA1001: Chlorambucil; Test type: Non-Inferiority or Equivalence — Comparability of dose-normalized PAAM Cmax values with ofatumumab in current study and without ofatumumab in prior study; Ratio of Cmax/Dose = 0.79, 90% CI 2-sided [0.63 to 0.99] — Ratio of Cmax/Dose is the ratio of dose-normalized PAAM Cmax values when given with ofatumumab in the current study and without ofatumumab in the prior study (LEUA1001)

18. Secondary Outcome: Dose-normalized AUC(0-6) and AUC(0-inf) of Chlorambucil and Dose-normalized AUC(0-6) of Phenylacetic Acid Mustard (PAAM)
Description: Blood samples for the determination of serum concentrations of chlorambucil and its metabolite PAAM were collected from participants in a substudy on Cycle 3 Day 1. The area under the plasma concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) and over 6 hours (AUC[0-6]) of chlorambucil and AUC(0-6) of PAAM normalized to the administered dose was determined as a measure of exposure and compared to reference data from a prior study (LEUA1001) [No NCT number available for this study; GlaxoSmithKline Document Number RM1998/00449/00].
Time Frame: Cycle 3 Day 1
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: Hours*nanogram/milliliter/milligram
Arm/Group | Study OMB110911: Ofatumumab + Chlorambucil | Study LEUA1001: Chlorambucil
Number analyzed (Participants) | 7 | 12
Hours*nanogram/milliliter/milligram
  Chlorambucil AUC(0-6)/Dose | 67.84 (0.24) | 65.43 (0.44)
  Chlorambucil AUC(0-inf)/Dose | 74.42 (0.23) | 67.10 (0.45)
  PAAM AUC(0-6)/Dose | 71.52 (0.26) | 80.32 (0.26)
Statistical Analysis 1: Comparison: Study OMB110911: Ofatumumab + Chlorambucil vs Study LEUA1001: Chlorambucil; Test type: Non-Inferiority or Equivalence — Comparability of dose-normalized chlorambucil AUC(0-6) values with ofatumumab in current study and without ofatumumab in prior study; Ratio of AUC(0-6)/Dose = 1.04, 90% CI 2-sided [0.77 to 1.40] — Ratio of AUC(0-6)/Dose is the ratio of dose-normalized chlorambucil AUC(0-6) values when given with ofatumumab in the current study and without ofatumumab in the prior study (LEUA1001)
Statistical Analysis 2: Comparison: Study OMB110911: Ofatumumab + Chlorambucil vs Study LEUA1001: Chlorambucil; Test type: Non-Inferiority or Equivalence — Comparability of dose-normalized chlorambucil AUC(0-inf) values with ofatumumab in current study and without ofatumumab in prior study; Ratio of AUC(0-inf)/Dose = 1.11, 90% CI 2-sided [0.82 to 1.50] — Ratio of AUC(0-inf)/Dose is the ratio of dose-normalized chlorambucil AUC(0-inf) values when given with ofatumumab in the current study and without ofatumumab in the prior study (LEUA1001)
Statistical Analysis 3: Comparison: Study OMB110911: Ofatumumab + Chlorambucil vs Study LEUA1001: Chlorambucil; Test type: Non-Inferiority or Equivalence — Comparability of dose-normalized PAAM AUC(0-6) values with ofatumumab in current study and without ofatumumab in prior study; Ratio of AUC(0-6)/Dose = 0.89, 90% CI 2-sided [0.72 to 1.10] — Ratio of AUC(0-6)/Dose is the ratio of dose-normalized PAAM AUC(0-6) values when given with ofatumumab in the current study and without ofatumumab in the prior study (LEUA1001)

19. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQOL)
Description: HRQOL was assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTCQLQC30), Chronic Lymphocytic Leukemia module (EORTC QLQ-CLL16), EuorQoL-Five Dimension (EQ-5D), and HCQ. Period (P)1 (Day 85, Day 169, Day 253) and P2 (scheduled follow-up (FU) and withdrawal visits) analysis were considered. Baseline (BL) for P1 was defined as score from screening visit and BL for P2 was defined as the last on-treatment score. The 2 principal QoL outcomes were pre-specified as the Global Health scale (GHS/QOL) of the EORTC QLQ-C30 and fatigue scale of the EORTC QLQ-CLL16. For EORTC QLQ-C30,GHS/Qol, the possible scale range was 0-100 (with 100 being 'best') and a positive difference from BL is indicative of better functioning (range -100 to +100). For the EORTC QLQ-CLL16 fatigue scale, the possible scale range was 0-100 (with 0 being 'best') and a negative difference from BL represents an improvement in fatigue (range -100 to +100).
Time Frame: Baseline, Cycle 4 day 1, cycle 7 day 1, 1 month follow-up, 6 month follow-up, 12 month follow-up
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 226 | 221
Scores on a scale
  P1, Cycle 4 Day 1, QLQC30 GHS/QoL score, n=139,159: number analyzed (Participants) | 139 | 159
  P1, Cycle 4 Day 1, QLQC30 GHS/QoL score, n=139,159 | 1.92 (21.22) | 6.08 (21.08)
  P1, Cycle 7 Day 1, QLQC30 GHS/QoL score, n=52, 55: number analyzed (Participants) | 52 | 55
  P1, Cycle 7 Day 1, QLQC30 GHS/QoL score, n=52, 55 | 8.01 (22.20) | 6.97 (17.55)
  P1,Cycle 4 Day 1,QLQCLL16 fatigue score, n=145,163: number analyzed (Participants) | 145 | 163
  P1,Cycle 4 Day 1,QLQCLL16 fatigue score, n=145,163 | -4.71 (27.48) | -4.60 (24.23)
  P1, Cycle 7 Day 1,QLQCLL16 fatigue score, n=55,57: number analyzed (Participants) | 55 | 57
  P1, Cycle 7 Day 1,QLQCLL16 fatigue score, n=55,57 | -1.21 (25.43) | -9.36 (22.93)
  P2,1 month FU, QLQC30 GHS/QoL score, n=118, 150: number analyzed (Participants) | 118 | 150
  P2,1 month FU, QLQC30 GHS/QoL score, n=118, 150 | 4.79 (23.13) | 0.56 (18.31)
  P2, 6 month FU, QLQC30 GHS/QoL score, n=83, 129: number analyzed (Participants) | 83 | 129
  P2, 6 month FU, QLQC30 GHS/QoL score, n=83, 129 | 3.01 (22.07) | 3.75 (20.83)
  P2, 12 month FU, QLQC30 GHS/QoL score, n=48, 96: number analyzed (Participants) | 48 | 96
  P2, 12 month FU, QLQC30 GHS/QoL score, n=48, 96 | 3.82 (18.27) | 1.22 (17.69)
  P2, 1 month FU, QLQCLL16 fatigue score, n=121, 152: number analyzed (Participants) | 121 | 152
  P2, 1 month FU, QLQCLL16 fatigue score, n=121, 152 | -1.24 (21.75) | -0.33 (19.13)
  P2, 6 month FU, QLQCLL16 fatigue score, n=85, 131: number analyzed (Participants) | 85 | 131
  P2, 6 month FU, QLQCLL16 fatigue score, n=85, 131 | -7.06 (18.96) | -2.93 (19.34)
  P2, 12 month FU, QLQCLL16 fatigue score, n=51, 95: number analyzed (Participants) | 51 | 95
  P2, 12 month FU, QLQCLL16 fatigue score, n=51, 95 | -2.94 (17.86) | 0.88 (16.91)

20. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the first dose of study medication to 60 days after the last dose of study medication and until follow-up for SAEs unless initiation of subsequent anti-CLL therapy, up to approximately 111 months.
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants
  Any AE | 205 | 208
  Any SAE | 84 | 97

21. Secondary Outcome: Number of Participants With AEs and SAEs of Maximum Severity of Grade 3 or Higher
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs. Maximum severity grades were evaluated according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: as for outcome 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants
  Any AE, Grade 3 | 54 | 67
  Any AE, Grade 4 | 31 | 36
  Any AE, Grade 5 | 25 | 36
  Any SAE, Grade 3 | 36 | 34
  Any SAE, Grade 4 | 13 | 19
  Any SAE, Grade 5 | 25 | 36

22. Secondary Outcome: Number of Participants With at Least One Grade 3/Grade 4 Myelosuppression (Anemia, Neutropenia, and Thrombocytopenia)
Description: Participants with a Grade 3 or Grade 4 myelosuppression (anemia, neutropenia, and thrombocytopenia) are presented by treatment cycle. Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. AEs were graded according to NCI common terminology criteria for adverse events (CTCAE) grade, version 3.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: as for outcome 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants | 92 | 83

23. Secondary Outcome: Number of Participants With Autoimmune Hemolytic Anaemia (AIHA) Disease
Description: AIHA is a disease where the body's immune system fails to recognize red blood cells as "self" and begins destroying these red blood cells. The number of participants diagnosed with AIHA are presented.
Time Frame: as for outcome 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants | 6 | 4

24. Secondary Outcome: Number of Participants Who Received no Transfusion or at Least One Transfusion During the Study
Description: Participants who received no transfusion and at least one transfusion during the study are presented. Participants who took any blood products are counted in this table.
Time Frame: From start of treatment to the last study visit/withdrawal visit (Median follow-up approximately 28.9 months)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 217
Participants
  No transfusions | 159 | 168
  At least one transfusion | 68 | 49

25. Secondary Outcome: Mean Change From Baseline in the Immunoglobulin (Ig) Antibodies IgA, IgG, and IgM
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants. Baseline IgA, IgG, and IgM values are the last pre-dose assessment values performed on Cycle 1 Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: From start of treatment up to 30 days after last treatment
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Chlorambucil | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 227 | 221
Gram per liter
  IgA, n=175, 186: number analyzed (Participants) | 175 | 186
  IgA, n=175, 186 | 0.047 (0.5706) | 0.048 (0.4257)
  IgG, n=175, 186: number analyzed (Participants) | 175 | 186
  IgG, n=175, 186 | -0.458 (3.6177) | -0.268 (2.5430)
  IgM n=175, 186: number analyzed (Participants) | 175 | 186
  IgM n=175, 186 | -0.398 (4.7864) | -0.031 (0.2507)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 111 months
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 111 months.
Groups:
- Ofatumumab 1000 mg + Chlorambucil: Participants with CLL received intravenous (IV) infusions of ofatumumab on Day 1 (300 mg) and Day 8 (1000 mg) in the first cycle, followed by IV infusions of 1000 mg on the first day of each subsequent 28-day cycle in combination with chlorambucil 10 mg/m^2 orally on Days 1-7 of every 28-day cycle for a minimum of 3 cycles until best response or a maximum of 12 cycles.
- Total: All patients.
Arm/Group | Chlorambucil | Ofatumumab 1000 mg + Chlorambucil | Total
All-Cause Mortality (participants affected / at risk) | 99/227 | 84/217 | 183/444
Serious Adverse Events (participants affected / at risk) | 57/227 | 53/217 | 110/444
Other Adverse Events (participants affected / at risk) | 175/227 | 183/217 | 358/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorambucil (N=227) | Ofatumumab 1000 mg + Chlorambucil (N=217) | Total (N=444)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 8
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 8
Haemolysis (Blood and lymphatic system disorders) | 1 | 1 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Inflammation (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 5 | 6
Vascular stent restenosis (General disorders) | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Empyema (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Haemophilus infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 3 | 4
Lung infection (Infections and infestations) | 0 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 2 | 5
Oral herpes (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 1 | 2
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 11 | 8 | 19
Pneumonia legionella (Infections and infestations) | 1 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 2 | 2
Septic shock (Infections and infestations) | 1 | 1 | 2
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 1
Mycobacterium test (Investigations) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebellar ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 2
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 2
Tremor (Nervous system disorders) | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorambucil (N=227) | Ofatumumab 1000 mg + Chlorambucil (N=217) | Total (N=444)
Anaemia (Blood and lymphatic system disorders) | 27 | 16 | 43
Leukopenia (Blood and lymphatic system disorders) | 4 | 14 | 18
Neutropenia (Blood and lymphatic system disorders) | 36 | 57 | 93
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 30 | 86
Abdominal pain upper (Gastrointestinal disorders) | 5 | 11 | 16
Constipation (Gastrointestinal disorders) | 13 | 10 | 23
Diarrhoea (Gastrointestinal disorders) | 31 | 38 | 69
Nausea (Gastrointestinal disorders) | 57 | 43 | 100
Vomiting (Gastrointestinal disorders) | 24 | 23 | 47
Asthenia (General disorders) | 11 | 18 | 29
Chills (General disorders) | 1 | 18 | 19
Fatigue (General disorders) | 40 | 35 | 75
Oedema peripheral (General disorders) | 12 | 15 | 27
Pyrexia (General disorders) | 18 | 36 | 54
Bronchitis (Infections and infestations) | 10 | 11 | 21
Nasopharyngitis (Infections and infestations) | 19 | 9 | 28
Upper respiratory tract infection (Infections and infestations) | 16 | 12 | 28
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 17 | 17
Decreased appetite (Metabolism and nutrition disorders) | 20 | 13 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 11 | 23
Dizziness (Nervous system disorders) | 15 | 10 | 25
Headache (Nervous system disorders) | 7 | 18 | 25
Insomnia (Psychiatric disorders) | 17 | 12 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 33 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 25 | 35
Erythema (Skin and subcutaneous tissue disorders) | 2 | 11 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 12 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 26 | 37
Rash (Skin and subcutaneous tissue disorders) | 21 | 53 | 74
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 22 | 24
Flushing (Vascular disorders) | 1 | 11 | 12
Hypertension (Vascular disorders) | 1 | 11 | 12
Hypotension (Vascular disorders) | 2 | 12 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.